CLINICAL TRIAL: NCT01153893
Title: Safety, Reactogenicity and Immunogenicity Study of GSK Biologicals' Pneumococcal Vaccine GSK1024850A, Given Either as a Booster Dose or as a 2-dose Catch-up Immunization in Healthy Nigerian Children
Brief Title: Immunization of Children Previously Primed With GSK Pneumococcal Vaccine GSK1024850A and of Unprimed Children in Nigeria
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 113199
Record Dates: First submitted 2010-06-29; First posted 2010-06-30 (Estimated); Results first posted 2012-03-15 (Estimated); Last update posted 2018-09-20 (Actual); Status verified 2016-09

CONDITIONS: Infections, Streptococcal
Keywords: Pneumococcal disease; Pneumococcal vaccine; Catch-up vaccination; Immunogenicity; Booster vaccination; Safety
MeSH Terms: conditions — Streptococcal Infections; Pneumococcal Infections | interventions — Pentetic Acid

ARMS (2):
- Synflorix/Infanrix primed Group (Experimental): Subjects previously primed with the Synflorix™ vaccine in the primary study 110521 (NCT00678301) received a booster dose of the Synflorix™ vaccine co-administered with a booster dose of the Infanrix™ vaccine at 15-21 months of age. Synflorix™ vaccine was administered intramuscularly in the right thigh or deltoid muscle of the arm. Infanrix™ vaccine was administered intramuscularly in the left thigh or deltoid muscle of the arm.
  Interventions: Biological: Pneumococcal vaccine GSK1024850A; Biological: InfanrixTM
- Synflorix/Infanrix unprimed Group (Experimental): Unprimed subjects from the primary study 110521 (NCT00678301), not previously vaccinated with any pneumococcal vaccine, received a 2-dose catch-up vaccination of Synflorix™ vaccine at 15-21 and 17-23 months of age and a booster dose of Infanrix™ vaccine co-administered with the first dose of Synflorix™ vaccine at 15-21 months of age. Synflorix™ vaccine was administered intramuscularly in the right thigh or deltoid muscle of the arm. Infanrix™ vaccine was administered intramuscularly in the left thigh or deltoid muscle of the arm.
  Interventions: Biological: Pneumococcal vaccine GSK1024850A; Biological: InfanrixTM

INTERVENTIONS:
Biological: Pneumococcal vaccine GSK1024850A — Intramuscular injection, 1 or 2 doses
Biological: InfanrixTM — Intramuscular injection, 1dose
  Other Names: DTPa

SUMMARY:
The purpose of this trial is to assess the safety, reactogenicity and immunogenicity of GSK Biologicals' pneumococcal conjugate vaccine GSK1024850A when administered either as a booster dose or as a two dose catch-up vaccination in the second year of life to the Nigerian subjects previously enrolled in the primary vaccination study NCT00678301.

This protocol posting deals with objectives & outcome measures of the booster phase. The objectives & outcome measures of the primary phase are presented in a separate protocol posting (NCT number = NCT00678301).

ELIGIBILITY:
Inclusion Criteria:

* Subjects who the investigator believes that their parent(s)/Legally Acceptable Representative(s) (LAR(s)) can and will comply with the requirements of the protocol.
* A male or female, between and including 15-21 months of age at the time of visit 1.
* For the Pn-Pn group, subjects who completed the full vaccination course in study NCT00678301. For the Zil-Pn group, subjects who were previously enrolled in the control group of study NCT00678301.
* Written informed consent, signed or thumb printed, obtained from the parent(s)/LAR(s) of the subject. Where parent(s)/LAR(s) are illiterate, the consent form will be countersigned by a witness.
* Healthy subjects as established by medical history and clinical examination before entering into the study.

Exclusion Criteria:

* Use of any investigational or non-registered product other than the study vaccine(s)/product(s) within 30 days preceding the first dose of vaccine, or planned use during the study period.
* Chronic administration of immunosuppressants or other immune-modifying drugs within six months prior to vaccination.
* Planned administration/administration of a vaccine not foreseen by the study protocol during the period starting from 30 days before each dose of study vaccine and ending 30 days after. Locally recommended vaccines for example Oral Polio Vaccine or influenza vaccine are always allowed, even if concomitantly administered with the study vaccines, but should be documented in the CRF.
* Concurrently participating in another clinical study at any time during the study period, in which the subject has been or will be exposed to an investigational or a non-investigational product.
* Administration of any pneumococcal vaccine since the end of study NCT00678301.
* Any confirmed or suspected immunosuppressive or immunodeficient condition, since the end of study NCT00678301, based on medical history and physical examination.
* Major congenital defects or serious chronic illness.
* History of any progressive neurological disorders or seizures.
* Acute disease and/or fever at the time of enrolment.
* History of any reaction or hypersensitivity likely to be exacerbated by any component of the vaccines.
* Administration of immunoglobulins and/or any blood products less than 3 months prior to visit 1 or planned use during the study.
* Child in care.

Ages: 15 Months to 21 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 105 (Actual)
Dates: Start 2010-10-04; Primary Completion 2011-02-16 (Actual); Study Completion 2011-02-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Ikeja / Lagos, Nigeria

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- [Derived] Odusanya OO, Kuyinu YA, Kehinde OA, Shafi F, Francois N, Yarzabal JP, Dobbelaere K, Ruggeberg JU, Borys D, Schuerman L. Safety and immunogenicity of 10-valent pneumococcal nontypeable Haemophilus influenzae protein D conjugate vaccine (PHiD-CV) in Nigerian children: Booster dose and 2-dose catch-up regimens in the second year of life. Hum Vaccin Immunother. 2014;10(3):757-66. doi: 10.4161/hv.27276. Epub 2013 Dec 4. PMID 24356787
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Statistical Analysis Plan: 113199 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 113199 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 113199 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 113199 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 113199 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 113199 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The duration of the study depends on the group allocation. The duration of the study per subject can vary from 1 month (Synflorix/Infanrix primed Group) to 3 months (Synflorix/Infanrix unprimed Group).
Pre-assignment Details: Because of an issue with the informed consent of a child, the data of the child, who had a non-related to study medication serious adverse event, are not detailed in this analysis. Data were reanalyzed for the 104 subjects with data available.
Groups:
- Synflorix/Infanrix Primed Group: Subjects previously primed with the Synflorix™ vaccine in the primary study NCT00678301 received a booster dose of the Synflorix™ vaccine co-administered with a booster dose of the Infanrix™ vaccine at 15-21 months of age. Synflorix™ vaccine was administered intramuscularly in the right thigh or deltoid muscle of the arm. Infanrix™ vaccine was administered intramuscularly in the left thigh or deltoid muscle of the arm.
- Synflorix/Infanrix Unprimed Group: Unprimed subjects from the primary study NCT00678301, not previously vaccinated with any pneumococcal vaccine, received a 2-dose catch-up vaccination of Synflorix™ vaccine at 15-21 and 17-23 months of age and a booster dose of Infanrix™ vaccine co-administered with the first dose of Synflorix™ vaccine at 15-21 months of age. Synflorix™ vaccine was administered intramuscularly in the right thigh or deltoid muscle of the arm. Infanrix™ vaccine was administered intramuscularly in the left thigh or deltoid muscle of the arm.
Period: Overall Study
Arm/Group | Synflorix/Infanrix Primed Group | Synflorix/Infanrix Unprimed Group
Started | 68 (Issues with the informed consent obtained from one child led to related data not used in this report) | 36
Completed | 67 (Number of subjects who completed the follow-up visit at Month 1.) | 36 (Number of subjects who completed the follow-up visit at Month 3.)
Not Completed | 1 | 0
Not completed — Adverse Event | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Synflorix/Infanrix Primed Group | Synflorix/Infanrix Unprimed Group | Total
Number analyzed (Participants) | 68 | 36 | 104
Age, Continuous [Mean (Standard Deviation); unit: Months] | 16.7 (1.00) | 16.4 (0.91) | 16.55 (0.955)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 29 | 17 | 46
  Male | 39 | 19 | 58

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects Reporting Grade 3 Symptoms (Solicited and Unsolicited).
Description: Grade 3 symptom = severe symptom that prevented normal activity.
  Solicited local symptoms assessed were pain, redness and swelling.
  Solicited general symptoms assessed were drowsiness, fever, irritability and loss of appetite.
  Unsolicited AEs = Any AE reported in addition to those solicited during the clinical study. Also any "solicited" symptom with onset outside the specified period of follow-up for solicited symptoms was reported as an unsolicited adverse event.
Time Frame: Within 31 days (Day 0 to Day 30) after administration of a booster dose of Synflorix vaccine in the Synflorix/Infanrix primed Group.
Population: The Total Vaccinated cohort included all vaccinated subjects.
Measure: Count of Participants; unit: Participants
Arm/Group | Synflorix/Infanrix Primed Group | Synflorix/Infanrix Unprimed Group
Number analyzed (Participants) | 68 | 0
Participants
  Any symptom | 3 |
  General symptoms | 1 |
  Local symptoms | 2 |

2. Secondary Outcome: Concentrations of Antibodies Against Vaccine Pneumococcal Serotypes.
Description: Vaccine pneumococcal serotypes assessed were serotypes 1, 4, 5, 6B, 7F, 9V, 14, 18C, 19F and 23F.
  Concentrations were expressed as geometric mean concentrations (GMCs) in microgram per millilitre (µg/mL).
  Pneumococcal serotype specific total imunoglobuline G (IgG) antibodies were measured by 22F-inhibition Enzyme-linked immunosorbent assay (ELISA). The cut-off of the assay was 0.05 µg/mL.
Time Frame: Prior to and one month after the booster immunisation for the Synflorix/Infanrix primed Group and prior to the first dose and one month after Dose 2 in the Synflorix/Infanrix unprimed Group
Population: The According-To-Protocol cohort for immunogenicity included all evaluable subjects for whom immunogenicity data were available. This included subjects for whom assay results were available for antibodies against at least one pneumococcal vaccine serotype or protein D for the blood sample taken one month after vaccination.
Measure: Geometric Mean (95% Confidence Interval); unit: µg/mL
Arm/Group | Synflorix/Infanrix Primed Group | Synflorix/Infanrix Unprimed Group
Number analyzed (Participants) | 68 | 35
µg/mL
  Anti-1 [pre-booster;pre-vacc] | 0.29 [0.22 to 0.40] | 0.03 [0.03 to 0.04]
  Anti-1 [post-booster;post-dose 2]: number analyzed (Participants) | 67 | 35
  Anti-1 [post-booster;post-dose 2] | 8.72 [6.37 to 11.93] | 3.17 [2.58 to 3.89]
  Anti-4 [pre-booster;pre-vacc] | 0.40 [0.31 to 0.50] | 0.06 [0.04 to 0.09]
  Anti-4 [post-booster;post-dose 2]: number analyzed (Participants) | 67 | 35
  Anti-4 [post-booster;post-dose 2] | 11.03 [9.06 to 13.42] | 8.22 [6.75 to 10.02]
  Anti-5 [pre-booster;pre-vacc] | 0.49 [0.40 to 0.61] | 0.05 [0.04 to 0.07]
  Anti-5 [post-booster;post-dose 2]: number analyzed (Participants) | 67 | 35
  Anti-5 [post-booster;post-dose 2] | 10.34 [8.32 to 12.85] | 2.87 [2.22 to 3.71]
  Anti-6B [pre-booster;pre-vacc] | 0.63 [0.48 to 0.83] | 0.05 [0.03 to 0.08]
  Anti-6B [post-booster;post-dose 2]: number analyzed (Participants) | 67 | 35
  Anti-6B [post-booster;post-dose 2] | 4.31 [3.37 to 5.52] | 0.85 [0.52 to 1.38]
  Anti-7F [pre-booster;pre-vacc] | 0.73 [0.57 to 0.92] | 0.05 [0.04 to 0.08]
  Anti-7F [post-booster;post-dose 2]: number analyzed (Participants) | 67 | 35
  Anti-7F [post-booster;post-dose 2] | 10.30 [8.57 to 12.38] | 6.07 [4.89 to 7.52]
  Anti-9V [pre-booster;pre-vacc]: number analyzed (Participants) | 67 | 35
  Anti-9V [pre-booster;pre-vacc] | 1.04 [0.78 to 1.39] | 0.06 [0.04 to 0.10]
  Anti-9V [post-booster;post-dose 2]: number analyzed (Participants) | 67 | 35
  Anti-9V [post-booster;post-dose 2] | 11.49 [9.02 to 14.65] | 2.70 [2.05 to 3.55]
  Anti-14 [pre-booster;pre-vacc] | 1.13 [0.87 to 1.46] | 0.14 [0.08 to 0.23]
  Anti-14 [post-booster;post-dose 2]: number analyzed (Participants) | 67 | 35
  Anti-14 [post-booster;post-dose 2] | 14.14 [11.74 to 17.04] | 10.59 [8.70 to 12.89]
  Anti-18C [pre-booster;pre-vacc] | 1.62 [1.30 to 2.04] | 0.05 [0.03 to 0.09]
  Anti-18C [post-booster;post-dose 2]: number analyzed (Participants) | 67 | 35
  Anti-18C [post-booster;post-dose 2] | 35.33 [27.73 to 45.02] | 25.61 [19.70 to 33.30]
  Anti-19F [pre-booster;pre-vacc]: number analyzed (Participants) | 67 | 35
  Anti-19F [pre-booster;pre-vacc] | 1.20 [0.85 to 1.71] | 0.14 [0.08 to 0.24]
  Anti-19F [post-booster;post-dose 2]: number analyzed (Participants) | 67 | 35
  Anti-19F [post-booster;post-dose 2] | 9.26 [7.20 to 11.91] | 7.16 [4.27 to 12.02]
  Anti-23F [pre-booster;pre-vacc] | 0.46 [0.32 to 0.68] | 0.03 [0.02 to 0.04]
  Anti-23F [post-booster;post-dose 2]: number analyzed (Participants) | 67 | 35
  Anti-23F [post-booster;post-dose 2] | 6.99 [5.21 to 9.39] | 1.06 [0.66 to 1.70]

3. Secondary Outcome: Concentrations of Antibodies Against Cross-reactive Pneumococcal Serotypes.
Description: Cross-reactive pneumococcal serotypes assessed were serotypes 6A and 19A. Concentrations were expressed as geometric mean concentrations (GMCs) in microgram per millilitre (µg/mL).
  The antibody concentrations against the cross-reactive pneumococcal serotypes 6A and 19A were determined by 22F-inhibition Enzyme-linked immunosorbent assay (ELISA). The cut-off of the assay was 0.05 µg/mL.
Time Frame: as for outcome 2
Population: as for outcome 2
Measure: Geometric Mean (95% Confidence Interval); unit: µg/mL
Arm/Group | Synflorix/Infanrix Primed Group | Synflorix/Infanrix Unprimed Group
Number analyzed (Participants) | 68 | 35
µg/mL
  Anti-6A [pre-booster;pre-vacc] | 0.19 [0.13 to 0.27] | 0.05 [0.03 to 0.07]
  Anti-6A [post-booster;post-dose 2]: number analyzed (Participants) | 67 | 35
  Anti-6A [post-booster;post-dose 2] | 0.81 [0.56 to 1.18] | 0.24 [0.15 to 0.40]
  Anti-19A [pre-booster;pre-vacc] | 0.24 [0.17 to 0.36] | 0.09 [0.05 to 0.17]
  Anti-19A [post-booster;post-dose 2]: number analyzed (Participants) | 67 | 35
  Anti-19A [post-booster;post-dose 2] | 1.33 [0.88 to 2.00] | 1.94 [1.13 to 3.33]

4. Secondary Outcome: Opsonophagocytic Activity Against Vaccine Pneumococcal Serotypes.
Description: Vaccine pneumococcal serotypes assessed were serotypes 1, 4, 5, 6B, 7F, 9V, 14, 18C, 19F and 23F.
  Streptococcus pneumoniae opsonophagocytic activity was measured by a killing-assay using a HL 60 cell line. The results were presented as the dilution of serum (opsonic titre) able to sustain 50% killing of live pneumococci under the assay conditions. The cut-off of the assay is an opsonic titre of 8.
Time Frame: One month after the booster immunisation for the Synflorix/Infanrix primed Group and one month after Dose 2 in the Synflorix/Infanrix unprimed Group
Population: as for outcome 2
Measure: Geometric Mean (95% Confidence Interval); unit: Titres
Arm/Group | Synflorix/Infanrix Primed Group | Synflorix/Infanrix Unprimed Group
Number analyzed (Participants) | 67 | 35
Titres
  Opsono-1 [post-booster;post-dose 2]: number analyzed (Participants) | 66 | 35
  Opsono-1 [post-booster;post-dose 2] | 1667.8 [1210.9 to 2297.0] | 103.4 [67.7 to 157.9]
  Opsono-4 [post-booster;post-dose 2]: number analyzed (Participants) | 65 | 35
  Opsono-4 [post-booster;post-dose 2] | 3869.1 [3122.8 to 4793.9] | 1482.9 [1211.0 to 1815.8]
  Opsono-5 [post-booster;post-dose 2] | 679.9 [515.9 to 895.9] | 58.7 [38.6 to 89.4]
  Opsono-6B [post-booster;post-dose 2]: number analyzed (Participants) | 66 | 31
  Opsono-6B [post-booster;post-dose 2] | 1687.6 [1138.7 to 2501.0] | 325.7 [118.1 to 898.6]
  Opsono-7F [post-booster;post-dose 2] | 11045.3 [8456.8 to 14426.3] | 7980.2 [6287.8 to 10128.1]
  Opsono-9V [post-booster;post-dose 2]: number analyzed (Participants) | 66 | 35
  Opsono-9V [post-booster;post-dose 2] | 5300.1 [4329.3 to 6488.5] | 6375.3 [4779.4 to 8504.1]
  Opsono-14 [post-booster;post-dose 2]: number analyzed (Participants) | 66 | 35
  Opsono-14 [post-booster;post-dose 2] | 2472.0 [1767.3 to 3457.8] | 1797.8 [1241.4 to 2603.6]
  Opsono-18C [post-booster;post-dose 2] | 2323.0 [1403.1 to 3846.1] | 4104.2 [2954.5 to 5701.2]
  Opsono-19F [post-booster;post-dose 2]: number analyzed (Participants) | 65 | 34
  Opsono-19F [post-booster;post-dose 2] | 683.5 [440.0 to 1062.0] | 443.5 [203.0 to 968.8]
  Opsono-23F [post-booster;post-dose 2] | 5144.5 [3657.4 to 7236.3] | 3081.7 [1389.3 to 6836.1]

5. Secondary Outcome: Opsonophagocytic Activity Against Cross-reactive Pneumococcal Serotypes.
Description: Cross-reactive pneumococcal serotypes assessed were serotypes 6A and 19A.
  Streptococcus pneumoniae opsonophagocytic activity was measured by a killing-assay using a HL 60 cell line. The results were presented as the dilution of serum (opsonic titre) able to sustain 50% killing of live pneumococci under the assay conditions. The cut-off of the assay is an opsonic titre of 8.
Time Frame: as for outcome 4
Population: as for outcome 2
Measure: Geometric Mean (95% Confidence Interval); unit: Titres
Arm/Group | Synflorix/Infanrix Primed Group | Synflorix/Infanrix Unprimed Group
Number analyzed (Participants) | 66 | 35
Titres
  Opsono-6A [post-booster;post-dose 2]: number analyzed (Participants) | 61 | 34
  Opsono-6A [post-booster;post-dose 2] | 213.0 [121.7 to 372.9] | 313.9 [147.6 to 667.4]
  Opsono-19A [post-booster;post-dose 2] | 112.7 [66.7 to 190.5] | 341.2 [159.0 to 732.1]

6. Secondary Outcome: Concentration of Antibodies Against Protein D (PD).
Description: Anti-PD antibodies were determined using an ELISA assay. Concentrations were expressed as geometric mean concentrations (GMCs) in ELISA units per millilitre (EL.U/mL). Concentration of specific PD antibodies was determined, using a standard reference serum. The cut-off of the assay is 100 ELISA units per millilitre (EL.U/mL).
Time Frame: as for outcome 2
Population: as for outcome 2
Measure: Geometric Mean (95% Confidence Interval); unit: EL.U/mL
Arm/Group | Synflorix/Infanrix Primed Group | Synflorix/Infanrix Unprimed Group
Number analyzed (Participants) | 67 | 35
EL.U/mL
  Anti-PD [pre-booster;pre-vacc]: number analyzed (Participants) | 66 | 35
  Anti-PD [pre-booster;pre-vacc] | 270.4 [211.7 to 345.3] | 61.5 [52.0 to 72.7]
  Anti-PD [post-booster;post-dose 2] | 2955.3 [2342.0 to 3729.2] | 501.1 [345.0 to 727.9]

7. Secondary Outcome: Number of Subjects Reporting Any and Grade 3 Solicited Local AEs.
Description: Solicited AEs = AEs to be recorded as endpoints in the clinical study. The presence/occurrence/intensity of these events was actively solicited from the subject or an observer during a specified post-vaccination follow-up period.
  Solicited local symptoms assessed were pain, redness and swelling.
  Any = occurrence of any local symptom regardless of intensity grade.
  Grade 3 pain = cried when limb was moved/spontaneously painful. Grade 3 redness/swelling = redness/swelling above 30 millimetre (mm)
Time Frame: Within 4 days (Days 0-3) after vaccination.
Population: The Total Vaccinated cohort included all vaccinated subjects.
Measure: Count of Participants; unit: Participants
Arm/Group | Synflorix/Infanrix Primed Group | Synflorix/Infanrix Unprimed Group
Number analyzed (Participants) | 68 | 36
Participants
  Any pain | 27 | 13
  Grade 3 pain | 0 | 0
  Any redness | 1 | 1
  Redness > 30 mm | 0 | 1
  Any swelling | 4 | 2
  Swelling > 30 mm | 2 | 1

8. Secondary Outcome: Number of Subjects Reporting Any, Grade 3 and Related Solicited General AEs.
Description: Solicited general symptoms assessed were drowsiness, irritability, loss of appetite and fever (= axillary temperature equal to or above 37.5 degrees Celsius (°C)).
  Any= occurrence of any general symptom regardless of intensity grade or relationship to vaccination Grade 3 drowsiness = drowsiness which prevented normal activity. Grade 3 irritability = crying that could not be comforted/ prevented normal activity. Grade 3 loss of appetite = not eating at all. Grade 3 fever = temperature >39.5°C.
  Related = solicited symptom assessed by the investigator as causally related to study vaccination.
Time Frame: Within 4 days (Days 0-3) after vaccination.
Population: The Total Vaccinated cohort included all vaccinated subjects.
Measure: Count of Participants; unit: Participants
Arm/Group | Synflorix/Infanrix Primed Group | Synflorix/Infanrix Unprimed Group
Number analyzed (Participants) | 68 | 36
Participants
  Any drowsiness | 2 | 0
  Grade 3 drowsiness | 0 | 0
  Related drowsiness | 2 | 0
  Fever >= 37.5°C | 8 | 3
  Fever > 39.5°C | 0 | 1
  Related fever | 8 | 3
  Any irritability | 2 | 0
  Grade 3 irritability | 0 | 0
  Related irritability | 2 | 0
  Any loss of appetite | 1 | 1
  Grade 3 loss of appetite | 0 | 0
  Related loss of appetite | 1 | 1

9. Secondary Outcome: Number of Subjects Reporting Unsolicited AEs.
Description: Unsolicited AEs = Any AE (i.e. any untoward medical occurrence in a patient or clinical investigation subject, temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product) reported in addition to those solicited during the clinical study. Also any "solicited" symptom with onset outside the specified period of follow-up for solicited symptoms was reported as an unsolicited adverse event.
Time Frame: Within 31 days (Days 0-30) after vaccination
Population: The Total Vaccinated cohort included all vaccinated subjects.
Measure: Count of Participants; unit: Participants
Arm/Group | Synflorix/Infanrix Primed Group | Synflorix/Infanrix Unprimed Group
Number analyzed (Participants) | 68 | 36
Participants | 31 | 18

10. Secondary Outcome: Number of Subjects Reporting Serious Adverse Events (SAEs).
Description: SAEs assessed include medical occurrences that results in death, are life threatening, require hospitalization or prolongation of hospitalization, results in disability/incapacity or are a congenital anomaly/birth defect in the offspring of a study subjects.
Time Frame: During the entire study period, from the vaccination visit at Day 0 up to the end of the follow-up visit at Month 1 for the Synflorix/Infanrix primed Group and up to Month 3 for the Synflorix/Infanrix unprimed Group.
Population: The Total Vaccinated cohort included all vaccinated subjects.
Measure: Count of Participants; unit: Participants
Arm/Group | Synflorix/Infanrix Primed Group | Synflorix/Infanrix Unprimed Group
Number analyzed (Participants) | 68 | 36
Participants | 1 | 0

ADVERSE EVENTS:
Time Frame: Solicited AEs: Within 4 days (Days 0-3) after vaccination. Unsolicited AEs: Within 31 days (Days 0-30) after vaccination. SAEs: From Day 0 up to Month 1 for the Synflorix/Infanrix primed Group and up to Month 3 for the Synflorix/Infanrix unprimed Group.
Description: Because of an issue discovered with the informed consent obtained for one child after the original statistical analysis. The data of the child, who also had an SAE that was not considered to be related to the study medication by the investigator, have been removed from the results tables.
Arm/Group | Synflorix/Infanrix Primed Group | Synflorix/Infanrix Unprimed Group
Serious Adverse Events (participants affected / at risk) | 1/68 | 0/36
Other Adverse Events (participants affected / at risk) | 46/68 | 25/36
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Synflorix/Infanrix Primed Group (N=68) | Synflorix/Infanrix Unprimed Group (N=36)
Drowning (General disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Synflorix/Infanrix Primed Group (N=68) | Synflorix/Infanrix Unprimed Group (N=36)
Respiratory tract infection (Infections and infestations) | 13 | 7
Malaria (Infections and infestations) | 8 | 10
Conjunctivitis (Eye disorders) | 3 | 2
Furuncle (Infections and infestations) | 4 | 1
Upper respiratory tract infection (Infections and infestations) | 3 | 2
Enteritis (Gastrointestinal disorders) | 0 | 2
Fever (General disorders) | 8 | 3
Pain (General disorders) | 27 | 13
Swelling (General disorders) | 4 | 2

LIMITATIONS AND CAVEATS:
Data were reanalyzed because an issue was discovered with the informed consent obtained for one child after the original statistical analysis. The child's parent requested GlaxoSmithKline not to use the data of their child.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.